CLINICAL TRIAL: NCT01340833
Title: Determination of the Absolute Bioavailability of GSK2118436 Following a Single Oral Dose Co-Administered With an Intravenous Radiolabelled Microtracer of GSK2118436 in Subjects With BRAF Mutant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113479
Record Dates: First submitted 2011-04-14; First posted 2011-04-25 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: GSK2118436; BRAF inhibitor; BRAF-mutation positive tumor; Oncology; absolute bioavailability; microtracer
MeSH Terms: conditions — Neoplasms | interventions — dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Medication (Experimental): GSK2118436
  Interventions: Drug: GSK2118436

INTERVENTIONS:
Drug: GSK2118436 — Two capsules each containing 75 mg GSK2118436, followed by a single IV dose of 50 ug (no more than 7.4 kBq or 200 nCi) [14C]GSK2118436, starting 1.75 hours after the oral dose

SUMMARY:
GSK2118436 is an orally administered, potent and selective small molecule BRAF inhibitor that is currently being developed for the treatment of BRAF mutation-positive tumors. This is an open-label, non-randomized study designed to determine the absolute bioavailability of an oral dose of 150 mg of GSK2118436 co-administered with an intravenous 50 microgram dose of [14C]GSK2118436 in subjects with BRAF mutant solid tumors. Pharmacokinetic samples will be obtained up to 72 hours post-dose. Safety assessments will be performed throughout the study. After completing all assessments, eligible subjects may transition to BRF114144, an open-label, rollover study of GSK2118436 to continue treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age at the time of signing the informed consent form;
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form;
* Body weight >/= 45 kg and a body mass index >/= 19 kg/m2 and </= 35 kg/m2 (inclusive);
* Able to swallow and retain oral medication;
* BRAF mutation-positive tumor as determined via relevant genetic testing;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Women of child-bearing potential and men with reproductive potential must be willing to practice acceptable methods of birth control. Additionally, women of childbearing potential must have a negative serum pregnancy test within 14 days prior to the first dose of study treatment;
* Must have adequate organ function as defined by the following values:

ANC >/=1.2 x 109/L Hemoglobin >/=9 g/dL Platelets >/=100 x 109/L Serum bilirubin </=1.5 x upper limit of normal (ULN) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) </= 2.5 x ULN; <5 x ULN if liver metastases are present Serum creatinine </= ULN or calculated creatinine clearance >/= 60 mL/min Prothrombin time / INR and partial thromboplastin time </=1.3 x ULN Left ventricular ejection fraction >/= institutional lower limit of normal by ECHO

Exclusion Criteria:

* Currently receiving cancer therapy (e.g., chemotherapy with delayed toxicity, extensive radiation therapy, immunotherapy, biologic therapy) within the last 3 weeks; chemotherapy regimens without delayed toxicity within the last 2 weeks; or use of an investigational anti-cancer drug within 28 days preceding the first dose of GSK2118436; use of any other investigational product within 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is warranted by data);
* Has participated in a 14C human research study in the 12 months prior to administration of study medication;
* Current use of a prohibited medication or requires any of these medications during the study;
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication;
* Current use of therapeutic warfarin (note: low molecular weight heparin and prophylactic low-dose warfarin are permitted);
* History of sensitivity to heparin or heparin-induced thrombocytopenia;
* Any major surgery within the last 4 weeks;
* Unresolved toxicity greater than National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (NCI CTCAE v4.0) [NCI, 2009] Grade 2 from previous anti-cancer therapy except alopecia;
* Presence of active gastrointestinal disease or other condition (e.g., small bowel or large bowel resection) that will interfere significantly with the absorption of drugs. If clarification is needed as to whether a condition will significantly affect absorption of drugs, contact the GSK medical monitor for permission to enrol the subject;
* A history of known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (subjects with documented laboratory evidence of HBV clearance may be enrolled);
* Presence of invasive malignancy other than one of the malignancies covered under Inclusion Criterion; subjects with a history of another malignancy that has been definitively treated can be enrolled;
* Subjects with brain metastases are excluded if their brain metastases are either:

Symptomatic Treated (surgery, radiation therapy), but not clinically and radiographically stable for a period of at least one month prior to study entry, or Asymptomatic and untreated but > 1 cm in the longest dimension Exception: Subjects with small (≤ 1 cm in the longest dimension), asymptomatic brain metastases that do not need immediate local therapy can be enrolled. Subjects on a stable dose of corticosteroids for more than one month, or those who have been off corticosteroids for at least 2 weeks can be enrolled. Subjects must also be off of enzyme-inducing anticonvulsants for more than 4 weeks;

* Corrected QT (QTc) interval >/= 480 msecs;
* History of acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting within the past 24 weeks;
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system; abnormal cardiac valve morphology documented by ECHO [subjects with minimal abnormalities (i.e., mild regurgitation/stenosis) can be entered on study - if clarification is needed as to whether an ECHO abnormality is minimal, please contact the GSK medical monitor); or history of known cardiac arrhythmias (except sinus arrythmias) within the past 24 weeks;
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drugs, or excipients (note: to date there are no known drugs chemically related to GSK2118436 which are approved by the FDA);
* Uncontrolled medical conditions (e.g., diabetes mellitus, hypertension), psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol; or history of alcohol or drug abuse within 6 months prior to screening; or unwillingness or inability to follow the procedures required in the protocol;
* Subjects with known glucose 6 phosphate dehydrogenase (G6PD) deficiency;
* Donation of blood or blood products in excess of 500 mL within the 56 days prior to administration of study medication;
* Pregnant females as determined by positive β hCG test at screening or prior to dosing or lactating females who are actively breast feeding;
* Subject is mentally or legally incapacitated;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-06-08 (Actual); Primary Completion 2011-09-12 (Actual); Study Completion 2011-09-12 (Actual)

PRIMARY OUTCOMES:
The percent of absolute bioavailability (F) of GSK2118436 following single-dose oral HPMC capsule and a concomitant IV microdose | Up to 72 hours

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of plasma GSK2118436 and [14C]GSK2118436 | Up to 72 hours
Time to Cmax (Tmax) of plasma GSK2118436 and [14C]GSK2118436 | Up to 72 hours
Area under the plasma-concentration time curve (AUC) of plasma GSK2118436 and [14C]GSK2118436 | Up to 72 hours
Terminal half-life (t1/2) of plasma GSK2118436 and [14C]GSK2118436 | Up to 72 hours
Oral clearance (CL/F) of GSK2118436 | Up to 72 hours
Clearance (CL) of [14C]GSK2118436 | Up to 72 hours
Volume of distribution (Vd) of [14C]GSK2118436 | Up to 72 hours
Number of subjects with adverse events as a measure of safety and tolerability | From date of dosing until transition to rollover protocol BRF114144 (approximately 4 days) or study follow up visit if subject does not transition to BRF114144 (approximately 11 - 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tacoma, Washington, United States

REFERENCES:
- [Background] Denton CL, Minthorn E, Carson SW, Young GC, Richards-Peterson LE, Botbyl J, Han C, Morrison RA, Blackman SC, Ouellet D. Concomitant oral and intravenous pharmacokinetics of dabrafenib, a BRAF inhibitor, in patients with BRAF V600 mutation-positive solid tumors. J Clin Pharmacol. 2013 Sep;53(9):955-61. doi: 10.1002/jcph.127. Epub 2013 Jul 12. PMID 23846776
- See also: Results for study 113479 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113479?search=study&search_terms=113479#rs